CLINICAL TRIAL: NCT02900781
Title: Comparative Effectiveness of an Activity-specific Monitoring Device- StepRite - on Short Term Outcomes in Adults After Partial or Total Knee Arthroplasty
Brief Title: Comparative Effectiveness of an Activity-specific Monitoring Device- StepRite
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants were unable to use the device. No data was collected
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: MedHab, LC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: L16-138
Record Dates: First submitted 2016-08-23; First posted 2016-09-14 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis; Degenerative Joint Disease
Keywords: Arthroplasty; Physical Therapy
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator Steprite™ Device' (Active Comparator): steprite™ device active Comparator- The steprite™ System is a monitoring and biofeedback system for the Monitoring of rehabilitation patients Measuring pressure distribution, gait and range of motion of the lower extremities while a patient performs specified rehabilitation exercises
  Interventions: Device: Steprite™
- Control (Placebo Comparator): Control outcomes with no device. Standard of care physical therapy and outcomes.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Steprite™ — Steprite™ Device shoe insert monitoring device
  Other Names: steprite™ System Device
  Arms: Active Comparator Steprite™ Device'
Other: Standard of care — No Device. Standard of care physical therapy
  Arms: Control

SUMMARY:
Partial or Total Knee Arthroplasty are procedures commonly used in severe degeneration of the knee joint due to osteoarthritis. With an increasing number of Partial or Total Knee Arthroplasty performed in a population that is aging during a time where the amount of healthcare dollars allotted to rehabilitation is declining, there is a need to develop remote monitoring of rehabilitation and to engage and optimize self-management of recovery.

Current management of Partial or Total Knee Arthroplasty recovery is typically performed in the out-patient setting and is highly protocol driven. A typical case might be seen by the physical therapist 2-3x/week for 8-10 weeks to perform specific exercises and to monitor progress (i.e. compliance with ROM and strengthening exercises). One recent study suggested that variation in patients' independent exercise and activity after arthroplasty surgery may contribute to variable functional gains.

The investigators are proposing that the StepRite device developed by MedHab, (a shoe insert that collects functional data) will reduce cost and improve the efficacy of rehabilitation in total knee arthroplasty patients

DETAILED DESCRIPTION:
Significance of this study The significance of the proposed study includes the projected benefit to the patients in terms of attaining clinical outcomes quicker and to the medical system in terms of managing cost for the provision of services. Subjects are expected to demonstrate improved compliance to patient tailored rehabilitation protocols which will lead to more rapid attainment of clinical outcomes versus present traditional rehabilitation methodologies. The expected level of, and rate of, attainment of clinical outcomes will translate to an overall reduction of cost to the medical system by reducing the need to engage in additional processes or the need to protract the time required to attain clinical outcomes, where either or both in combination can increase rehabilitation expenditures.

Objectives To compare the efficacy of StepRite in a prescribed physical therapy program verses traditional in-facility physical therapy program after partial or total knee replacement surgery using validated survey tools to evaluate patient progress, including patient self -reporting of progress and surgeon appraisal of patient performance post-operatively.

To compare the overall cost of post-operative rehabilitation of patients involved in traditionally employed regimens versus those using the StepRite device.

Hypothesis and specific aims The aim of this study is to evaluate whether improved clinical outcomes as well as reduction in cost in provision of care can be better affected through the use of the Steprite device as compared to the use of traditional rehabilitation modalities.

The Investigators will seek to reject the null hypotheses that 1) there is no difference between clinical outcomes attained between patients using the Steprite device and those using traditional rehabilitation modalities and that 2) there is no reduction in cost to the medical system when patients use Steprite versus other conventional methods of rehabilitation.

By rejecting the null hypothesis the investigators will accept the alternate hypothesis that, through the use of the Steprite device, not only will patients achieve overall clinical outcomes faster but there will be an associated decrease in cost burden to the medical system and the differences observed will be statistically significant as compared to rehabilitation of patients not using the Steprite device.

Patients who use the device post-surgery will demonstrate superior short-term improvements (i.e. 3 months post surgery) with respect to self-reported functional outcomes and gait parameters, compared to a control group not using the device. The patients will self-report through the use of validated survey instruments including the KOOS survey (knee injury and osteoarthritis outcome score), LEFS (lower extremity functional scale) and/or KSS (knee society score), the latter of which includes a section for surgeon evaluation of patient functionality post operatively.

Study Design and Methods This is a point of care clinical trial; a trial that functions to integrate research within a clinical setting that has the ability to readily deliver either modality of the proposal. This type of study design relies on provider referral of patients to be approached for consent, after which randomization to one of two treatment groups is facilitated; a control group of 15 patients participating in conventional rehabilitation regimens and an experimental group of 15 patients who will participate in the same rehabilitation regimen but facilitated through the use of Steprite. Importantly, care for patients is delivered as part of current adopted standards utilizing outcome measurements, the use of which and the interpretation of which is already built into care provided by the clinical facility, thereby negating the need to develop additional outcome measures.

Recruitment of 30 patients will come from the investigators' normal patient population, among patients who are scheduled for partial or total knee arthroplasty. As there is no change in post op care for these patients from the investigators standard protocols other than monitoring and enforcement of home protocols, the same therapists involved in investigators' normal patient care will be involved with both arms of the study.

For this study, 30 patients represents a sample size deemed acceptable as a starting point. There are no other published studies using Steprite in comparative design trials. Determinations of sample size needed for this study, using 80% power and significance of 0.05, incorporate the use of a time frame in days or weeks for completion of the rehabilitation protocols that would allow for the detection of clinically significant differences between the group using Steprite and those using conventional therapies only. Given that conventional therapies can include skilled nursing, home health and outpatient visits and given that the need for each of these is highly variable dependent on the patient, it is difficult to assign a time value for determinations of sample size.

With that, a sample size of 30 participants divided into two groups represents an initial starting point, with the potential of incremental addition of more patients in order to achieve significance between the two study groups.

Statistical significance will be evaluated utilizing a standard t-test for two group comparison.

In preparation for the study, MedHab Inc. will at their expense train all involved investigators and therapists in the fitting and use of the StepRite device. Medhab will also train a lead therapist designated by the lead investigator to be in charge of overseeing and monitoring, ensuring proper use of the device. There is no cost to the patient, hospital or other funding entity for participation in this study. Medhab LLC will assume all costs associated with the training, application, device and use of the StepRite product for the full course of this study.

Subjects for this study will be recruited from the patient population seen by the investigator's during the normal course of business. There will be no outside recruitment of individuals or advertising as to the presence or use of the monitoring device to entice new patient referral. Prospective candidates will be asked by the investigator at the time they are designated surgical candidates. All documentation related to the study will be reviewed with the patient by the lead physician or his designee who is appropriately trained in discussing patient recruitment. Final decision and randomization to control or StepRite use will be done as part of the preoperative checkup just prior to surgery where both operative consent and study consent are discussed and signed.

Randomization:

Once a patient agrees to the study they would be sequentially randomized into whether or not they receive StepRite. The patients will be randomized to every other eligible patient gets the intervention. (ie: 1,3,5,7,9… will get StepRite ; 2,4,6,8 will not get StepRite) 15 Intervention subjects will be recruited and 15 control subjects will be recruited with an extra 5 patients to account for attrition and withdrawals.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral partial or total knee arthroplasty.
* Age 45-75 yr. old
* BMI <35
* Access to Wi-Fi
* Have appropriate smart phone and knowledge of use
* Be willing to place StepRite app on their personal phone

Exclusion Criteria:

* History of neuromuscular disorder (e.g. Parkinson's, Polio, or stroke).
* Pregnancy
* History of cognitive disease that would preclude ability to navigate smart phone

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W Brindley, MD, Principal Investigator — TTUHSC
Locations (1):
- TTUHSC Orthopaedic Surgery MS 9436, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consented participants
Pre-assignment Details: StudyTerminated- device not working
Groups:
- Device: Device group- Standard of Care with the device
Period: Overall Study
Arm/Group | Control | Device
Started (Study terminated due to device not working at our facility .) | 4 | 5
Completed (Participants were unable to use the device as required in the protocol. No data collected) | 0 | 0
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Population: Study Terminated after 9 patients consented due to device not working at our site. No data was collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator Steprite™ Device' | Control | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Partial or Total Knee Arthroplasty [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Step Rite Device
Description: Effectiveness of outcomes with the use of the StepRite device
Time Frame: 3 months
Population: Study Terminated due to device not working at our site. No data collected
Groups:
- Control: control group
- StepRite Device: Device group
Arm/Group | Control | StepRite Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse event data was not collected due to the study being terminated. The device did not work and NO data was collected
Description: study Terminated. Unable to use device. No data collected
Groups:
- Device: Device group
Arm/Group | Control | Device
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT02900781/Prot_SAP_000.pdf